CLINICAL TRIAL: NCT01190449
Title: A Phase II Trial of Ofatumumab (CALGB IND #) in Previously Untreated Follicular Non-Hodgkin's Lymphoma (NHL)
Brief Title: Ofatumumab in Treating Patients With Previously Untreated Stage II, Stage III, or Stage IV Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50901; CALGB-50901; GSK-CALGB-50901; CDR0000683083 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive high-dose ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once monthly in months 3-9.
  Interventions: Biological: ofatumumab
- Arm II (Experimental): Patients receive a lower dose of ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once monthly in months 3-9.
  Interventions: Biological: ofatumumab

INTERVENTIONS:
Biological: ofatumumab — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as ofatumumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This randomized phase II trial is studying ofatumumab to see how well it works in treating patients with previously untreated stage II, stage III, or stage IV follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate in patients with previously untreated CD20-positive bulky stage II, or stage III or IV follicular non-Hodgkin lymphoma (NHL) treated with a lower- or high-dose of ofatumumab.

Secondary

* To determine the progression-free survival (PFS) of patients treated with these regimens.
* To determine the toxicity profile of these regimens in these patients.
* To establish whether the therapeutic effect of single-agent ofatumumab is sufficiently promising to warrant evaluation in subsequent randomized, ofatumumab-based, biologic doublet trials.
* To evaluate the two ofatumumab doses by independent comparison of response, PFS, and toxicity to a historical control in previously untreated patients with follicular NHL.
* To prospectively validate the FLIPI2 prognostic index in low- and intermediate-risk patients and compare to low- and intermediate-risk stratified patients by standard FLIPI scoring to determine a more reliable indicator of response and PFS.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive high-dose ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once monthly in months 3-9.
* Arm II: Patients receive a lower dose of ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once monthly in months 3-9.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients may undergo blood and bone marrow sample collection for correlative studies.

After completion of study therapy, patients are followed up every 4 months for 2 years and then every 6 months for 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular non-Hodgkin lymphoma (NHL) meeting 1 of the following criteria:

  * Bulky (i.e., single mass ≥ 7cm in any uni-dimensional measurement) stage II disease
  * Stage III or IV disease
* WHO grade 1, 2, or 3a disease
* Bone marrow biopsies allowed provided they are submitted in conjunction with nodal biopsies

  * No fine-needle aspirates for diagnosis
* Tumor tissue must express the CD20-positive antigen by flow cytometry or IHC
* At least 1 site of measurable disease that is > 1 cm in diameter in ≥ 1 dimension present either on physical exam or imaging studies

  * Non-measurable disease alone not allowed, including the following:

    * Bone lesions (lesions if present should be noted)
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Bone marrow (involvement by NHL should be noted)
* Low- or intermediate-risk disease by the Follicular Lymphoma International Prognostic Index (FLIPI)

  * FLIPI score meeting 1 or 2 of the following risk factors:

    * Age > 60 years
    * Involvement of > 4 nodal sites
    * Stage III-IV disease
    * Hemoglobin < 12.0 g/dL
    * LDH normal
  * Risk determined by the following:

    * Low Risk: 0-1 of the above risk factors
    * Intermediate Risk: 2 risk factors
    * Poor Risk: ≥ 3 risk factors
* No known CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Creatinine clearance ≥ 30 mL/min
* Bilirubin ≤ 2 times upper limit of normal (unless secondary to Gilbert syndrome or hepatic involvement of NHL)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Patients with HIV infection allowed provided the following criteria are met:

  * No evidence of coinfection with hepatitis B or C
  * CD4+ cell count ≥ 400/mm³
  * No evidence of resistant strains of HIV
  * HIV viral load < 10,000 copies HIV RNA/mL if not on anti-HIV therapy OR HIV viral load < 50 copies if on anti-HIV therapy
  * No history of AIDS-defining conditions
* No evidence of active hepatitis B (HBV) or C (HCV) infection (i.e., no positive serology for anti-HBc or anti-HCV antibodies)

  * HBV seropositivity allowed (HBsAg+) provided they are closely monitored for evidence of active HBV infection by HBV DNA testing
  * After completing treatment, HBsAg + patients must be monitored by HBV DNA testing every 2 months for 6 months post-treatment, while continuing lamivudine (required)

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or immunotherapy (e.g., monoclonal antibody-based therapy) for NHL

  * Prior involved-field radiation therapy allowed
* More than 2 weeks since prior corticosteroids except for maintenance therapy for a non-malignant disease

  * No concurrent dexamethasone or other steroids as antiemetics
* No live virus vaccination within 6 weeks prior to study entry
* No concurrent zidvoudine or stavudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cara A. Rosenbaum, MD, Principal Investigator — University of Chicago
Locations (48):
- United States (48):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - Union Hospital of Cecil County, Elkton, Maryland
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Mount Kisco Medical Group, PC, Mount Kisco, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Low-dose Ofatumumab): Patients receive a lower dose (500 mg) of ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once every 8 weeks in months 3-9 (weeks 12, 20, 28, and 36).
- Arm II (High-dose Ofatumumab): Patients receive a high-dose (1000 mg) of ofatumumab IV over 2-8 hours on days 1, 8, 15, and 22 and then once every 8 weeks in months 3-9 (weeks 12, 20, 28, and 36).
Period: Overall Study
Arm/Group | Arm I (Low-dose Ofatumumab) | Arm II (High-dose Ofatumumab)
Started | 15 | 36
Completed | 15 | 32
Not Completed | 0 | 4
Not completed — Ineligible | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics summarized overall for all patients who enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Low-dose Ofatumumab) | Arm II (High-dose Ofatumumab) | Total
Number analyzed (Participants) | 15 | 36 | 51
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 85] | 58 [40 to 85] | 60 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 19 | 23
  Male | 11 | 17 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 36 | 51

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Complete or Partial Response) by Month 12
Description: The primary endpoint of this trial is overall response rate (OR=complete response (CR) or partial response (PR)) to 500 mg or 1000 mg dose of ofatumumab in previously untreated patients with CD20+ follicular NHL. The response outcome is defined as the best response during the 12 months of first-line and extended induction treatment. A CR is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A PR is defined as at least a 50% decrease in the sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses, with no increase observed in the size of other nodes, liver, or spleen and no new sites of disease should be observed. The ORR (percentage of patients) reported below by arm is the percentage of patients whose best response during the 12 months of treatment was CR or PR.
Time Frame: From baseline to month 12
Population: Patients who completed the study and were not ineligible were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Low-dose Ofatumumab) | Arm II (High-dose Ofatumumab)
Number analyzed (Participants) | 15 | 32
percentage of patients | 60 [32 to 84] | 84 [67 to 95]

2. Secondary Outcome: Median Progression-free Survival Time
Description: The median progression-free survival (PFS) time for each arm was estimated using the Kaplan-Meier method. PFS was calculated as the time from study entry until progression or death, whichever occurred first. Patients were censored at the time last known alive and progression free. Lymph nodes should be considered abnormal if the long axis is > 1.5 cm, regardless of the short axis. If a lymph node has a long axis of 1.1 to 1.5 cm, it should only be considered abnormal if its short axis is > 1.0. Lymph nodes ≤ 1.0 cm by ≤ 1.0 cm will not be considered as abnormal for relapse or progressive disease. Progression is defined using the 2007 revised response criteria reported by Cheson et al. as follows: Appearance of any new lesion, At least a 50% increase from nadir in the SPD of any previously involved nodes, At least a 50% increase in the longest diameter of any single previously identified node > 1.0 cm in its short axis.
Time Frame: From date of study entry until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 4 years
Population: Patients who completed the study and were not ineligible were included in this analysis.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm I (Low-dose Ofatumumab) | Arm II (High-dose Ofatumumab)
Number analyzed (Participants) | 15 | 32
years | 1.9 [1.0 to 1.9] | 1.9 [1.5 to 3.0]

ADVERSE EVENTS:
Time Frame: From baseline to month 12
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed the study. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I (Low-dose Ofatumumab) | Arm II (High-dose Ofatumumab)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/15 | 8/36
Other Adverse Events (participants affected / at risk) | 15/15 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose Ofatumumab) (N=15) | Arm II (High-dose Ofatumumab) (N=36)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 3 (3)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose Ofatumumab) (N=15) | Arm II (High-dose Ofatumumab) (N=36)
Anemia (Blood and lymphatic system disorders) | 2 (5) | 6 (23)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (4) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (4)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (20)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (7)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (8)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (18)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (18)
Flatulence (Gastrointestinal disorders) | 1 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (7)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (8) | 13 (29)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 1 (1) | 4 (11)
Edema limbs (General disorders) | 1 (2) | 3 (10)
Edema trunk (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (32) | 23 (75)
Fever (General disorders) | 1 (1) | 4 (5)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 2 (2)
Infusion related reaction (General disorders) | 13 (19) | 29 (33)
Malaise (General disorders) | 0 (0) | 1 (1)
Neck edema (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (2) | 4 (9)
Allergic reaction (Immune system disorders) | 1 (3) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (2)
Bronchial infection (Infections and infestations) | 1 (1) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (7)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (11)
Creatinine increased (Investigations) | 1 (2) | 3 (5)
Lymphocyte count decreased (Investigations) | 3 (17) | 11 (41)
Neutrophil count decreased (Investigations) | 0 (0) | 6 (12)
Platelet count decreased (Investigations) | 2 (9) | 2 (11)
Weight gain (Investigations) | 1 (2) | 3 (7)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (5) | 10 (26)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (10) | 12 (46)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (7) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 6 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (16)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (12) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (6)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 5 (9)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (12) | 9 (19)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 3 (9)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (7) | 5 (16)
Confusion (Psychiatric disorders) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (11)
Insomnia (Psychiatric disorders) | 4 (6) | 11 (29)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (8)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 7 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 12 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (12)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (6)
Flushing (Vascular disorders) | 0 (0) | 2 (5)
Hot flashes (Vascular disorders) | 1 (2) | 2 (2)
Hypertension (Vascular disorders) | 3 (13) | 11 (45)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Lymphedema (Vascular disorders) | 0 (0) | 1 (2)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes